CLINICAL TRIAL: NCT02177812
Title: A Phase I Open-label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of GSK2879552 Given Orally in Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: A Phase I Dose Escalation Study of GSK2879552 in Subjects With Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The risk benefit in relapsed refractory AML does not favor continuation of the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200200
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-04

CONDITIONS: Leukaemia, Myelocytic, Acute
Keywords: Oncology; LSD1; GSK2879552; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Neoplasms; Leukemia, Myeloid, Acute | interventions — GSK2879552

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Escalation Phase (Part 1) (Experimental): The safety and PK/PD data will be reviewed prior to the dose decision, and the dose escalation will be guided by the Neuenschwander -continuous reassessment method (N-CRM).The dose escalation will complete when RP2D is determined. The RP2D will be the MTD or a lower dose that provides adequate PK exposure and biologic activity with superior tolerability.
  Interventions: Drug: GSK2879552; Drug: ATRA
- Expansion Phase (Part 2) (Experimental): Once the MTD and/or RP2D has been determined in Part 1, an expansion cohort of up to 30 subjects will be enrolled in order to characterize the clinical activity and safety profile of the RP2D. Subjects may continue treatment in the study until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: GSK2879552; Drug: ATRA

INTERVENTIONS:
Drug: GSK2879552 — GSK2879552 capsules contain 0.25 mg, 0.5 mg, 2 mg or 5 mg of GSK2879552 as parent. The initial dosing regimen will be continuous oral daily dosing.
Drug: ATRA — ATRA (Tretinoin) will be supplied as a 10 mg capsule for oral administration. The initial dosing regimen will be continuous oral twice daily dosing

SUMMARY:
This study is a phase I, open-label study to determine recommended phase 2 dose (RP2D) and regimen for the orally administered lysine specific demethylase 1 (LSD1) inhibitor GSK2879552, alone or in combination with All-Trans Retinoic Acid (ATRA). The recommended dose and regimen will be selected based on the safety, pharmacokinetic (PK), and pharmacodynamic (PD) profiles observed after the treatment of subjects with relapsed/refractory AML. The study consists of two parts. Part 1 will identify the maximum tolerated dose (MTD) and/or RP2D using a dose-escalation procedure. Dose escalations will be guided by the Neuenschwander-continual reassessment method (N-CRM). PK/PD expansion cohorts will also be included in Part 1 to characterize the range of biologically effective doses by assessing PD markers and obtain additional PK data. Part 2 will explore further the safety, tolerability, and clinical activity of GSK2879552, alone or in combination with ATRA, at the RP2D in subjects with AML.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >=18 years of age and provided signed written informed consent.
* Subjects must have relapsed/refractory AML by world health organization (WHO) classification for which no standard therapies are available or anticipated to result in a durable remission. French- American- British system (FAB) subtype M3 will be excluded.
* Subjects >= 60 years of age with AML who are not candidates for or have refused standard chemotherapy.
* Subjects who have previously received an autologous stem cell transplant are allowed if a minimum of 3 months has elapsed from the time of transplant and the subject has recovered from transplant-associated toxicities prior to the first dose of GSK2879552.
* Subjects with a history of allogeneic stem cell transplant are eligible for study participation provided the following eligibility criteria are met: transplant was >60 days prior to study enrolment; subject has not taken immunosuppressive medications for at least 1 month; no signs or symptoms of graft versus host disease other than Grade 1 skin involvement; no active infection.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Subjects must be stable and, in the opinion of the investigator, be expected to complete 4 week treatment period.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* All prior treatment-related toxicities must be National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 4.0 <=Grade 1 at the time of enrollment (except for alopecia).
* Adequate baseline organ function.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose of study treatment and agree to use effective contraception, during the study and for 7 days (GSK2879552 mono therapy) or 30 days (combination with ATRA), following the last dose of study treatment.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from the administration of the first dose of study treatment until 3 months after the last dose of study treatment to allow for clearance of any altered sperm.

Exclusion Criteria:

* Active human immunodeficiency virus (HIV), Hepatitis B Virus (HBV) or hepatitis C virus (HCV) infections at the time of screening. Subjects with laboratory evidence of HCV clearance may be enrolled.
* History of or concurrent malignancy of solid tumours, except: subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible. Subjects with second malignancies that are indolent or definitively treated may be enrolled even if less than 5 years have elapsed since treatment. Consult GlaxoSmithKline (GSK) Medical Monitor if unsure whether second malignancies meet requirements specified above.
* Currently receiving cancer therapy. Hydroxyurea will be allowed.
* Received major surgery, radiotherapy, or immunotherapy within 4 weeks of GSK2879552 administration.
* Prior treatment with temozolomide, dacarbazine or procarbazine
* Prior treatment with poly ADP ribose polymerase (PARP) inhibitors (eg., olaparib, ABT-888)
* Baseline Montreal Cognitive Assessment (MOCA) score of 22 or lower
* Evidence of severe or uncontrolled systemic diseases. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator
* Current active liver or biliary disease.
* Patients at risk of non-AML related major bleeding (e.g. recent gastrointestinal [GI] hemorrhage or neurosurgery).
* Symptomatic or untreated central nervous system (CNS) leukemia. Subjects are permitted to enroll if previously treated for CNS disease, free of symptoms at the time of screening, and have not required intrathecal chemotherapy at least 1 month prior to study Day 1.
* Cardiac abnormalities
* Administration of an investigational drug within 14 days or 5 half-lives, whichever is shorter with a minimum of 14 days preceding the first dose of study treatment(s) in this study.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK2879552 or LSD1 inhibitors that contraindicates their participation.
* Lactating female.
* Consumption of Seville oranges, grapefruit, grapefruit hybrids, grapefruit juice, pommelos, or exotic citrus fruits, from 1 day prior to the first dose of study treatment(s) until the last dose of study drug.
* Current use of a prohibited medication including anticoagulants or platelet inhibitors or expected to require any of these medications during treatment with the investigational drug.
* Previous treatment with GSK2879552 For ATRA Combination arm ONLY
* Known hypersensitivity to ATRA, parabens (preservatives in the gelatin capsule) or other retinoids.
* ATRA capsule contains sorbitol. Subjects with rare hereditary problems of fructose intolerance are excluded.
* History of seizure within 12 months or brain tumor (primary)
* History of taking mega-dose vitamin A (>25,000 USP U/day) within 3 months from the dosing start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (6):
- United States (4):
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Melbourne, Victoria, Australia
- GSK Investigational Site, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 41 participants with relapsed/refractory acute myeloid leukemia (AML) were enrolled in Part 1 at different centers in Australia, Canada and United States. This study was planned to be conducted in 2 parts :Part 1 (dose escalation) and Part 2 (Expansion Cohort).
Pre-assignment Details: This study was terminated early during Part 1 as the risk benefit in relapsed/refractory AML did not favor continuation of the study and therefore, Part 2 was not conducted. There were no active participants on study when the study was terminated.
Groups:
- Part 1:GSK2879552 1mg QD: Participants received GSK2879552 1 milligram (mg) orally once daily (QD) in fasted condition with approximately 200 milliliter (mL) of water
- Part 1: GSK2879552 2mg QD: Participants received GSK2879552 2 mg orally once daily in fasted condition with approximately 200 mL of water
- Part 1: GSK2879552 4mg QD: Participants received GSK2879552 4 mg orally once daily in fasted condition with approximately 200 mL of water.
- Part 1: GSK2879552 8mg QD: Participants received GSK2879552 8 mg orally once daily in fasted condition with approximately 200 mL of water
- Part 1: GSK2879552 12mg QD: Participants received GSK2879552 12 mg orally once daily in fasted condition with approximately 200 mL of water.
- Part 1: GSK2879552 20mg QD: Participants received GSK2879552 20 mg orally once daily in fasted condition with approximately 200 mL of water.
- Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day: Participants received GSK2879552 2 mg capsule orally once daily in fasted condition with approximately 200 mL of water in combination with All-Trans Retinoic Acid (ATRA) at a dose of 45 mg per meter square per day (mg/m^2/day).
- Part 1: GSK2879552 20mg QD PK/PD Expansion: Participants received GSK2879552 20 mg capsule orally once daily in fasted condition with approximately 200 mL of water in Pharmacokinetic/Pharmacodynamics (PK/PD) Expansion cohort to collect adequate data on safety, PK or PD.
- Part 2: Expansion Cohort: In Part 2, participants were planned to receive the recommended Phase 2 dose of GSK2879552 orally once daily in fasted condition with approximately 200 mL of water alone or in combination with ATRA
Period: Part 1 (Median of 4 Weeks)
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion | Part 2: Expansion Cohort
Started | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6 | 0
Completed | 1 | 2 | 7 | 4 | 5 | 1 | 1 | 4 | 0
Not Completed | 0 | 0 | 0 | 1 | 1 | 3 | 9 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 1 | 6 | 1 | 0
Period: Part 2 (Up to 14 Months)
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion | Part 2: Expansion Cohort
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was not collected for Part 2, as no participants were enrolled in Part 2.
Groups:
- Part 1:GSK2879552 1mg QD: Participants received GSK2879552 1 mg orally QD in fasted condition with approximately 200 mL of water.
- Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day: Participants received GSK2879552 2 mg capsule orally once daily in fasted condition with approximately 200 mL of water in combination with ATRA at a dose of 45 mg/m^2/day.
- Part 1: GSK2879552 20mg QD PK/PD Expansion: Participants received GSK2879552 20 mg capsule orally once daily in fasted condition with approximately 200 mL of water in PK/PD Expansion cohort to collect adequate data on safety, PK or PD.
- Total: Total of all reporting groups
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion | Part 2: Expansion Cohort | Total
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6 | 0 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (NA) — Standard Deviation could not be calculated as only one participant was analyzed | 73.5 (2.12) | 64.3 (5.77) | 61.0 (13.96) | 71.7 (4.08) | 71.8 (4.03) | 63.1 (20.14) | 65.5 (19.07) |  | 66.1 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 3 | 3 | 2 | 1 | 3 | 1 | 0 | 13
  Male | 1 | 2 | 4 | 2 | 4 | 3 | 7 | 5 | 0 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
  Asian - Central/South Asian Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Asian - East Asian Heritage | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 4
  Asian - South East Asian Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  White - White/Caucasian/European Heritage | 1 | 2 | 4 | 3 | 2 | 2 | 6 | 4 | 0 | 24
  Missing | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population comprised of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  All AEs | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
  All SAEs | 1 | 2 | 7 | 5 | 6 | 3 | 8 | 5

2. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLT)
Description: An event was considered a DLT if it occursed within the first 28 days of treatment, and meets one of the following criteria unless it can be clearly established that the event was unrelated to treatment: hematologic DLT included myelosuppression, Grade >=3 non-hematologic toxicity that is considered clinically significant and lasts >72 hours, Grade 2 toxicity that in the judgment of the investigator and GSK Medical Monitor is dose-limiting and treatment delay of >=42 days due to unresolved toxicity.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With AE Leading to Dose Reductions or Delays
Description: The number of participants who had any dose reduction or delay have been presented.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  AEs leading to dose reduction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  AEs leading to dose interruption/delay | 0 | 0 | 2 | 3 | 5 | 0 | 6 | 1

4. Primary Outcome: Part 1: Number of Participants With Withdrawals Due to Toxicities
Description: Participants were monitored from start of the study till the development of toxicity. The data for number of participants withdrawn due to toxicities has been presented.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants | 0 | 0 | 0 | 1 | 4 | 2 | 4 | 2

5. Primary Outcome: Number of Participants With Clinical Chemistry Parameters Changes From Baseline With Respect to the Normal Range
Description: Blood samples were collected to assess clinical chemistry parameters like urea/blood urea nitrogen (BUN), calcium, potassium, aspartate aminotransferase (AST), total bilirubin, direct bilirubin, creatinine, chloride, alanine aminotransferase (ALT), uric acid, glucose, total carbon dioxide (CO2), gamma glutamyl transferase (GGT), albumin, sodium, alkaline phosphatase, total protein, phosphate, lactate dehydrogenase (LDH). Laboratory values were as per local labs per site with own normal ranges. Values above range were reported as high and values below range as low. Data for worst case post Baseline is reported.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  Direct Bilirubin,to Low,n=1,2,7,5,6,4,10,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin,to High,n=1,2,7,5,6,4,10,6 | 0 | 0 | 2 | 1 | 2 | 0 | 5 | 3
  Chloride,to Low,n=1,2,7,5,6,4,10,6 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1
  Chloride,to High,n=1,2,7,5,6,4,10,6 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
  CO2/Bicarbonate,to Low,n=1,2,7,5,6,4,10,6 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 2
  CO2/Bicarbonate,to High,n=1,2,7,5,6,4,10,6 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1
  Lactate Dehydrogenase,to Low,n=1,2,7,5,6,4,10,6 | 0 | 0 | 2 | 2 | 2 | 0 | 2 | 2
  Lactate Dehydrogenase,to High,n=1,2,7,5,6,4,10,6 | 1 | 0 | 2 | 1 | 2 | 0 | 3 | 2
  Total Protein,to Low,n=1,2,7,4,6,4,10,6: number analyzed (Participants) | 1 | 2 | 7 | 4 | 6 | 4 | 10 | 6
  Total Protein,to Low,n=1,2,7,4,6,4,10,6 | 0 | 1 | 3 | 2 | 4 | 2 | 3 | 2
  Total Protein,to High,n=1,2,7,4,6,4,10,6: number analyzed (Participants) | 1 | 2 | 7 | 4 | 6 | 4 | 10 | 6
  Total Protein,to High,n=1,2,7,4,6,4,10,6 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  Urea/BUN,to Low,n=1,2,7,5,6,4,10,6 | 1 | 0 | 1 | 2 | 1 | 1 | 2 | 0
  Urea/BUN,to High,n=1,2,7,5,6,4,10,6 | 0 | 0 | 3 | 1 | 2 | 0 | 1 | 2

6. Primary Outcome: Number of Participants With Clinical Chemistry Toxicity Grade Changes From Baseline
Description: Blood samples were collected for analysis of clinical chemistry parameters based on common terminology criteria for adverse events (CTCAE) version 4.0, where Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe or medically significant; Grade 4 is life threatening consequences. Data for any increase in grade of worst-case on-therapy has been provided.
Time Frame: Median of 4 weeks of drug exposure
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  Albumin, n=1,2,7,5,6,4,10,6 | 1 | 2 | 5 | 3 | 4 | 4 | 6 | 3
  ALP, n=1,2,7,5,6,4, 10, 6 | 0 | 0 | 3 | 2 | 1 | 0 | 3 | 0
  ALT, n=1,2,7,5,6,4,10,6 | 0 | 0 | 4 | 3 | 1 | 1 | 5 | 2
  AST, n=1,2,7,5,6,4,10,6 | 1 | 2 | 3 | 2 | 1 | 1 | 3 | 1
  Total bilirubin, n=1,2,7,5,6,4,10,6 | 1 | 1 | 2 | 1 | 3 | 0 | 4 | 2
  Hypercalcemia, n=1,2,7,5,6,4,10,6 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0
  Hypoglycemia,n= 1,2,7,5,6,4,10,6 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0
  Creatinine,n=1,2,7,5,6,4,10,6 | 0 | 1 | 2 | 1 | 1 | 0 | 4 | 1
  GGT,n=1,2,7,5,3,1,8,3: number analyzed (Participants) | 1 | 2 | 7 | 5 | 3 | 1 | 8 | 3
  GGT,n=1,2,7,5,3,1,8,3 | 0 | 0 | 5 | 4 | 2 | 0 | 5 | 2
  Hyperglycemia,n= 0,1,7,5,6,4,9,6: number analyzed (Participants) | 0 | 1 | 7 | 5 | 6 | 4 | 9 | 6
  Hyperglycemia,n= 0,1,7,5,6,4,9,6 | 0 | 0 | 4 | 2 | 1 | 0 | 4 | 4
  Hypoglycemia,n=0,1,7,5,6,4,9,6: number analyzed (Participants) | 0 | 1 | 7 | 5 | 6 | 4 | 9 | 6
  Hypoglycemia,n=0,1,7,5,6,4,9,6 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hyperkalemia,n=1,2,7,5,6,4,10,6 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Hypokalemia,n=1,2,7,5,6,4,10,6 | 0 | 0 | 3 | 4 | 3 | 2 | 6 | 0
  Hypernatremia, n=1,2,7,5,6,4,10,6 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Hyponatremia, n=1,2,7,5,6,4,10,6 | 1 | 1 | 2 | 0 | 5 | 1 | 5 | 3
  Phosphorus, n=1,2,7,5,6,4,10,6 | 1 | 1 | 6 | 2 | 5 | 2 | 3 | 2

7. Primary Outcome: Number of Participants With Hematology Parameters Change From Baseline With Respect to the Normal Range
Description: Blood samples were collected to assess hematology parameters like mean corpuscle hemoglobin concentration (MCHC), mean corpuscle hemoglobin (MCH), mean corpuscle volume (MCV) mean platelet volume (MPV), basophils, eosinophils, hematocrit, hemoglobin, lymphocytes, monocytes, platelet count, Red blood cell (RBC) count, reticulocytes, White Blood Cell (WBC) count. Laboratory values were as per local labs per site with own normal ranges. Values above range were reported as high and values below range as low. Data for worst post Baseline were reported. NA indicates that data were not available as standard deviation could not be calculated for a single participant.
Time Frame: Median of 4 weeks of drug exposure
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  Basophils, to Low,n=1,2,7,4,2,2,9,5: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 9 | 5
  Basophils, to Low,n=1,2,7,4,2,2,9,5 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Basophils, to High,n=1,2,7,4,2,2,9,5: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 9 | 5
  Basophils, to High,n=1,2,7,4,2,2,9,5 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
  Eosinophils, to Low,n=1,2,7,4,2,2,8,5: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 8 | 5
  Eosinophils, to Low,n=1,2,7,4,2,2,8,5 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  Eosinophils, to High,n=1,2,7,4,2,2,8,5: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 8 | 5
  Eosinophils, to High,n=1,2,7,4,2,2,8,5 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Hemoglobin, to Low,n=0,0,0,0,2,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
  Hemoglobin, to Low,n=0,0,0,0,2,0,0,1 |  |  |  |  | 0 |  |  | 0
  Hemoglobin, to High,n=0,0,0,0,2,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
  Hemoglobin, to High,n=0,0,0,0,2,0,0,1 |  |  |  |  | 0 |  |  | 1
  Hematocrit, to Low,n=1,2,7,5,6,4,10,6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hematocrit, to High,n=1,2,7,5,6,4,10,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MCHC, to Low,n=1,2,7,5,3,2,10,6: number analyzed (Participants) | 1 | 2 | 7 | 5 | 3 | 2 | 10 | 6
  MCHC, to Low,n=1,2,7,5,3,2,10,6 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  MCHC, to High,n=1,2,7,5,3,2,10,6: number analyzed (Participants) | 1 | 2 | 7 | 5 | 3 | 2 | 10 | 6
  MCHC, to High,n=1,2,7,5,3,2,10,6 | 1 | 0 | 3 | 2 | 0 | 1 | 2 | 1
  MCH, to Low,n=1,2,7,5,3,2,10,6: number analyzed (Participants) | 1 | 2 | 7 | 5 | 3 | 2 | 10 | 6
  MCH, to Low,n=1,2,7,5,3,2,10,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MCH, to High,n=1,2,7,5,3,2,10,6: number analyzed (Participants) | 1 | 2 | 7 | 5 | 3 | 2 | 10 | 6
  MCH, to High,n=1,2,7,5,3,2,10,6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  MCV, to Low,n=1,2,7,5,6,4,10,6 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 2
  MCV, to High,n=1,2,7,5,6,4,10,6 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Monocytes, to Low,n=1,2,7,4,2,2,10,6: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 10 | 6
  Monocytes, to Low,n=1,2,7,4,2,2,10,6 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 1
  Monocytes, to High,n=1,2,7,4,2,2,10,6: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 10 | 6
  Monocytes, to High,n=1,2,7,4,2,2,10,6 | 0 | 1 | 4 | 0 | 1 | 1 | 2 | 2
  MPV, to Low,n=0,0,0,3,6,3,7,6: number analyzed (Participants) | 0 | 0 | 0 | 3 | 6 | 3 | 7 | 6
  MPV, to Low,n=0,0,0,3,6,3,7,6 |  |  |  | 1 | 1 | 1 | 0 | 1
  MPV, to High,n=0,0,0,3,6,3,7,6: number analyzed (Participants) | 0 | 0 | 0 | 3 | 6 | 3 | 7 | 6
  MPV, to High,n=0,0,0,3,6,3,7,6 |  |  |  | 1 | 2 | 0 | 3 | 4
  Nucleated RBC, to Low,n=0,0,0,1,1,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Nucleated RBC, to Low,n=0,0,0,1,1,0,1,0 |  |  |  | 0 | 0 |  | 0 |
  Nucleated RBC, to High,n=0,0,0,1,1,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Nucleated RBC, to High,n=0,0,0,1,1,0,1,0 |  |  |  | 0 | 0 |  | 0 |
  RBC, to Low,n=1,2,7,5,6,4,10,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC, to High,n=1,2,7,5,6,4,10,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reticulocytes, to Low,n=1,2,7,4,2,2,7,5: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 7 | 5
  Reticulocytes, to Low,n=1,2,7,4,2,2,7,5 | 0 | 2 | 5 | 1 | 2 | 1 | 2 | 1
  Reticulocytes, to High,n=1,2,7,4,2,2,7,5: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 7 | 5
  Reticulocytes, to High,n=1,2,7,4,2,2,7,5 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Hematology Toxicity Grade Changes From Baseline
Description: Blood samples were collected for analysis of hematology parameters based on common terminology criteria for adverse events (CTCAE) version 4.0, where Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe or medically significant; Grade 4 is life threatening consequences. Data for any grade increase worst-case on-therapy has been provided.
Time Frame: Median of 4 weeks of drug exposure
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  Hg increase,n=1,2,7,5,6,4,10,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hg anemia,n=1,2,7,5,6,4,10,6 | 1 | 2 | 5 | 4 | 1 | 2 | 4 | 3
  Lymph increase,n=1,2,7,4,2,2,10,6: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 10 | 6
  Lymph increase,n=1,2,7,4,2,2,10,6 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 1
  Lymph decrease,n=1,2,7,4,2,2,10,6: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 10 | 6
  Lymph decrease,n=1,2,7,4,2,2,10,6 | 1 | 2 | 2 | 3 | 1 | 2 | 5 | 2
  Total Neu,n=1,2,7,4,2,2,10,6: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 10 | 6
  Total Neu,n=1,2,7,4,2,2,10,6 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1
  Platelet,n=1,2,7,5,6,4,10,6 | 1 | 1 | 4 | 3 | 1 | 2 | 3 | 3
  WBC,n=1,2,7,5,6,4,10,6 | 1 | 2 | 2 | 4 | 5 | 1 | 5 | 1

9. Primary Outcome: Part 1: Number of Participants With Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured after resting for 5 minutes in semi-supine position. Vital signs were graded according to Common Toxicity Criteria for Adverse Events (CTCAE) version 4. An increase is defined as an increase in CTCAE grade relative to Baseline grade. For SBP Grade 0 (<120 millimeters of mercury [mmHg]), Grade 1 (120-139 mmHg), Grade 2 (140-159 mmHg), Grade 3 (>=160 mmHg). For DBP Grade 0 (<80 mmHg), Grade 1 (80-89 mmHg), Grade 2 (90-99 mmHg), Grade 3 (>=100 mmHg). Data for worst-case post Baseline is reported.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population. Only those participants with available data at the specified time points were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  SBP,Any Grade Increase; n=1, 1, 3, 4, 6, 2, 5, 3: number analyzed (Participants) | 1 | 1 | 3 | 4 | 6 | 2 | 5 | 3
  SBP,Any Grade Increase; n=1, 1, 3, 4, 6, 2, 5, 3 | 1 | 1 | 3 | 4 | 6 | 2 | 5 | 3
  SBP,Increase to Grade 2;n=1, 1, 3, 4, 6, 2, 5, 3: number analyzed (Participants) | 1 | 1 | 3 | 4 | 6 | 2 | 5 | 3
  SBP,Increase to Grade 2;n=1, 1, 3, 4, 6, 2, 5, 3 | 1 | 1 | 1 | 2 | 2 | 1 | 4 | 3
  SBP,Increase to Grade 3;n=1, 1, 3, 4, 6, 2, 5, 3: number analyzed (Participants) | 1 | 1 | 3 | 4 | 6 | 2 | 5 | 3
  SBP,Increase to Grade 3;n=1, 1, 3, 4, 6, 2, 5, 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
  DBP,Any Grade Increase;n=1, 2, 3, 2, 4, 1, 3, 2: number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 1 | 3 | 2
  DBP,Any Grade Increase;n=1, 2, 3, 2, 4, 1, 3, 2 | 1 | 2 | 3 | 2 | 4 | 1 | 3 | 2
  DBP,Increase to Grade 2;n=1, 2, 3, 2, 4, 1, 3, 2: number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 1 | 3 | 2
  DBP,Increase to Grade 2;n=1, 2, 3, 2, 4, 1, 3, 2 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 0
  DBP,Increase to Grade 3;n=1, 2, 3, 2, 4, 1, 3, 2: number analyzed (Participants) | 1 | 2 | 3 | 2 | 4 | 1 | 3 | 2
  DBP,Increase to Grade 3;n=1, 2, 3, 2, 4, 1, 3, 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Part 1: Number of Participants With Change From Baseline in Heart Rate
Description: Heart rate was measured after restings for 5 minutes in semi-supine position. Data for participants with heart rate decreased to < 60 beats per minute (bpm), normal or no change, increase to > 100 bpm. Data for worst post Baseline were reported.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  Decrease to <60 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Change to Normal or No Change | 0 | 2 | 1 | 4 | 4 | 4 | 5 | 3
  Increase to >100 | 1 | 0 | 6 | 1 | 2 | 0 | 5 | 3

11. Primary Outcome: Part 1: Number of Participants With Change From Baseline in Temperature
Description: Temperature was measured after resting for 5 minutes in semi-supine position. Data for participants with temperature decreased to <=35 Celsius, normal or no change, increase to >=38 Celsius at worst-case post Baseline is reported.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  Decrease to <=35 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Change to Normal or No Change | 1 | 2 | 4 | 4 | 5 | 4 | 9 | 6
  Increase to >=38 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0

12. Primary Outcome: Part 1: Number of Participants With Change From Baseline in Respiratory Rate
Description: Respiration rate was measured after resting for 5 minutes in semi-supine position. Data for worst case post-Baseline has been reported. Number of participants with respiratory rate decrease to <12 and increase to >25 has been reported.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  Decrease to <12 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Increase to >25 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0

13. Primary Outcome: Part 1: Number of Participants With Abnormal Electrocardiograms (ECGs) Findings
Description: A single 12-lead ECG was performed in semi-recumbent or supine position after 5 minutes of rest for the participant. An ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and corrected QT intervals was used. Number of participants with any visit post-Baseline abnormal clinically significant findings and abnormal not clinically significant findings in ECG results has been reported.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Participants
  Abnormal - not clinically significant | 1 | 2 | 7 | 4 | 4 | 2 | 4 | 6
  Abnormal - clinically significant | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1

14. Primary Outcome: Part 1: Number of Participants With Abnormal Physical Examinations
Description: Data for participants with abnormal physical examinations parameters was planned to be recorded.
Time Frame: Median of 4 weeks of drug exposure
Population: All Treated Subjects Population. The data was not collected as it was not captured within the case report form (CRF).
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Part 2: Objective Response Rate of Participants
Description: Objective response rate defined as the percentage of participants who achievied complete remission (CR), partial remission (PR), CRp (as per CR but platelet count <100 x 10^9/L) and morphologic leukemia free state per response criteria. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: All Treated Subjects Population. Data for this endpoint was not collected as this study was terminated early during Part 1 as the risk benefit in relapsed/refractory AML did not favor continuation of the study
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

16. Secondary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration [AUC(0-t)] and From Time Zero (Pre-dose) Extrapolated to Infinite Time [(AUC(0-inf)] After Single Dose Administration
Description: Blood samples were collected at indicated time points. The Pharmacokinetic (PK) parameters were calculated by non-compartmental analysis. NA indicates that data were not available as geometric co-efficient of variation could not be calculated for a single participant.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1
Population: PK Population comprised of all treated participants for whom a PK sample was obtained and analyzed. Only those participants with available data at the specified time points were analyzed (represented by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Hour*nanograms per milliliter
  AUC(0-t) n=1, 2, 7, 5, 6,4, 9,5: number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 9 | 5
  AUC(0-t) n=1, 2, 7, 5, 6,4, 9,5 | 30.9457 (NA) — NA indicates that data were not available as geometric co-efficient could not be calculated for a single participant. | 62.7579 (40.6) | 211.1387 (34.8) | 549.9557 (64.3) | 738.1552 (77.6) | 974.7759 (24.2) | 97.6341 (38.8) | 968.7825 (36.1)
  AUC(0-inf); n=1, 2, 7, 5, 6,4, 8,5: number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 8 | 5
  AUC(0-inf); n=1, 2, 7, 5, 6,4, 8,5 | 36.8470 (NA) — NA indicates that data were not available as geometric co-efficient could not be calculated for a single participant. | 72.7180 (31.4) | 222.0837 (35.1) | 600.6492 (61.9) | 791.2295 (74.1) | 1125.8508 (29.7) | 105.4513 (41.7) | 1101.4318 (41.0)

17. Secondary Outcome: Part 1: AUC Over the Dosing Interval (0-tau) After Single Dose Administration
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis. NA indicates that data were not available as geometric co-efficient could not be calculated for a single participant.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1
Population: PK Population. Only those participants with available data at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 8 | 5
Hour*nanograms per milliliter | 22.2630 (NA) — NA indicates that data were not available as geometric coefficient of variation could not be calculated for a single participant. | 44.0692 (45.5) | 169.5072 (35.1) | 483.7209 (62.2) | 638.4389 (70.3) | 870.8045 (21.0) | 80.2478 (48.4) | 885.8174 (24.1)

18. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration [AUC(0-t)] and AUC Over the Dosing Interval (0-tau) After Repeated Administration
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis. NA indicates that data were not available as geometric coefficient of variation could not be calculated for a single participant.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 15
Population: PK Population. Only those participants with available data at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 4 | 4 | 6 | 2 | 6 | 4
Hour*nanograms per milliliter
  AUC (0-t) | 22.0069 (NA) — NA indicates that data were not available as geometric coefficient of variation could not be calculated for a single participant. | 82.6381 (31.2) | 221.5336 (48.2) | 692.8434 (62.3) | 623.2032 (63.9) | 1158.6530 (27.3) | 132.0625 (38.4) | 904.0276 (30.2)
  AUC (0-tau) | 37.6629 (NA) — NA indicates that data were not available as geometric coefficient of variation could not be calculated for a single participant. | 82.8980 (31.5) | 221.6595 (48.2) | 699.1461 (62.3) | 661.7915 (58.0) | 1152.0895 (24.9) | 142.6193 (35.0) | 904.2889 (30.0)

19. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of GSK2879552
Description: as for outcome 18
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1 and 15
Population: PK Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Nanograms per milliliter
  Day 1,n=1,2,7,5,6,4,9,5: number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 9 | 5
  Day 1,n=1,2,7,5,6,4,9,5 | 4.0660 (NA) — NA indicates that data were not available as geometric coefficient of variation could not be calculated for a single participant. | 7.5501 (34.2) | 28.5460 (32.0) | 65.5650 (59.8) | 98.6033 (73.1) | 134.8388 (12.8) | 13.3889 (63.3) | 142.8826 (28.6)
  Day 15,n=1,2,4,4,6,2,6,4: number analyzed (Participants) | 1 | 2 | 4 | 4 | 6 | 2 | 6 | 4
  Day 15,n=1,2,4,4,6,2,6,4 | 4.3920 (NA) — NA indicates that data were not available as geometric coefficient of variation could not be calculated for a single participant. | 11.5411 (60.1) | 40.1989 (52.0) | 83.2978 (32.9) | 103.0141 (65.7) | 224.2444 (17.7) | 16.7684 (37.0) | 144.6871 (25.4)

20. Secondary Outcome: Part 1: Apparent Terminal Phase Half-life (t½)
Description: as for outcome 18
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1 and 15
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 8 | 5
Hours | 34.6647 (NA) — NA indicates that data were not available as geometric coefficient of variation could not be calculated for a single participant. | 29.7715 (37.3) | 19.6564 (15.9) | 11.2045 (26.0) | 12.4020 (26.5) | 15.9502 (20.6) | 14.9631 (38.9) | 10.5340 (47.8)

21. Secondary Outcome: Part 1: Time of Occurrence of Cmax (Tmax) of GSK2879552
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis. NA indicates that data were not available as standard deviation could not be calculated for a single participant.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1 and 15
Population: as for outcome 19
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Hours
  Day 1, n=1, 2, 7, 5, 6, 4, 9, 5: number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 9 | 5
  Day 1, n=1, 2, 7, 5, 6, 4, 9, 5 | 0.983 [0.983 to 0.983] | 0.7500 [0.500 to 1.000] | 1.0000 [0.500 to 2.000] | 0.9667 [0.467 to 1.500] | 1.2750 [0.500 to 2.500] | 0.6667 [0.500 to 1.033] | 1.0000 [0.333 to 1.750] | 1.0000 [0.500 to 1.000]
  Day 15, n= 1, 2, 4, 4, 6, 2, 6, 4: number analyzed (Participants) | 1 | 2 | 4 | 4 | 6 | 2 | 6 | 4
  Day 15, n= 1, 2, 4, 4, 6, 2, 6, 4 | 1.0000 [1.000 to 1.000] | 1.0000 [0.500 to 1.500] | 0.7833 [0.500 to 2.017] | 1.5833 [0.500 to 1.983] | 0.8167 [0.500 to 3.050] | 0.3833 [0.267 to 0.500] | 0.9917 [0.500 to 3.033] | 1.3000 [0.500 to 2.000]

22. Secondary Outcome: Part 1: Accumulation Ratio for GSK2879552
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis. Accumulation ratio was determined dividing AUC (0-tau) on Day 15 by AUC (0-tau) on Day 1. The ratio of accumulation of GSK2879552 was estimated by calculating the ratio of the geometric least squares (GLS) means of the AUC(0-tau) between Day 15 and Day 1 for all dose levels and the corresponding 90 percent confidence interval (CI) for each ratio.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1 and 15
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 2 | 4 | 4 | 6 | 2 | 6 | 4
Ratio | 1.881 [1.072 to 3.300] | 1.367 [1.208 to 1.547] | 1.319 [1.099 to 1.584] | 1.037 [0.792 to 1.356] | 1.388 [0.900 to 2.141] | 1.750 [1.449 to 2.113] | 1.073 [0.860 to 1.338]

23. Secondary Outcome: Part 1:Time Invariance
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis. The time invariance of GSK2879552 was estimated by calculating the ratio of the GLS means of the AUC (0-tau) between Day 15 and Day 1 for all dose levels and the corresponding 90 percent CI for each ratio.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1 and 15
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 0 | 2 | 4 | 4 | 6 | 2 | 6 | 4
Ratio |  | 1.140 [1.136 to 1.144] | 1.030 [0.891 to 1.191] | 1.042 [0.874 to 1.242] | 0.836 [0.657 to 1.065] | 1.167 [0.639 to 2.130] | 1.346 [1.164 to 1.556] | 0.845 [0.625 to 1.143]

24. Secondary Outcome: Part 1:Percentage of Participants With Objective Response
Description: Objective response rate is defined as the percentage of participants who achieved CR, PR, as per CR but platelet count <100 x 10^9/L and morphologic leukemia free state per response criteria.
Time Frame: Median of 4 weeks drug response
Population: All Treated Subjects.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion
Number analyzed (Participants) | 1 | 2 | 7 | 5 | 6 | 4 | 10 | 6
Percentage of Participants | 0 [0.0 to 97.5] | 0 [0.0 to 84.2] | 0 [0.0 to 41.0] | 0 [0.0 to 52.2] | 17 [0.4 to 64.1] | 0 [0.0 to 60.2] | 10 [0.3 to 44.5] | 0 [0.0 to 45.9]

25. Secondary Outcome: Part 1: AUC(0-t), AUC (0-tau) and AUC(0-inf) of ATRA
Description: Blood samples were collected at indicated time points. The Pharmacokinetic (PK) parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1and Day 15
Population: PK Population. Plasma samples were not quantifiable for ATRA at all end points and hence the PK parameters could not be derived.
Arm/Group | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day
Number analyzed (Participants) | 0

26. Secondary Outcome: Part 1: Cmax of ATRA
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1 and 15
Population: as for outcome 25
Arm/Group | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day
Number analyzed (Participants) | 0

27. Secondary Outcome: Part 1: Apparent Terminal Phase Half-life (t½) of ATRA
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1 and 15
Population: as for outcome 25
Arm/Group | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day
Number analyzed (Participants) | 0

28. Secondary Outcome: Part 1: Time of Occurrence of Cmax (Tmax) of ATRA
Description: Blood samples were collected at indicated time points. The PK parameters were calculated by non-compartmental analysis.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Day 1 and 15
Population: as for outcome 25
Arm/Group | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day
Number analyzed (Participants) | 0

29. Secondary Outcome: Part 2: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 15
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

30. Secondary Outcome: Part 2: Number of Participants With AE Leading to Dose Reductions or Delays
Description: The number of participants who had any dose reduction or delay have been presented. All dose reductions were due to AEs. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 15
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

31. Secondary Outcome: Part 2: Number of Participants With Withdrawals Due to Toxicities
Description: Participants were monitored from start of the study till the development of toxicity. The data for number of participants withdrawn due to toxicities has been presented. This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 15
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

32. Secondary Outcome: Part 2: Number of Participants With Abnormal Clinical Chemistry Parameters
Description: Data was not collected for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 15
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

33. Secondary Outcome: Part 2: Number of Participants With Abnormal Hematology Parameters
Description: Data was not collected for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 15
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

34. Secondary Outcome: Part 2: Number of Participants With Abnormal Vital Signs
Description: Data was not collected for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 15
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

35. Secondary Outcome: Part 2: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 15
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

36. Secondary Outcome: Part 2: Number of Participants With Abnormal Physical Examinations
Description: This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 15
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

37. Secondary Outcome: Part 2: Clearance (CL) of GSK2879552 for Part 2
Description: This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Day 1 (pre-dose, 0.5 and 3 hours post dose), Days 4, 8 (pre-dose), Day 15 (pre-dose, 0.5, 1, 4, 6 hours), Weeks 4, 5, 6, 7, 8 and every 4 weeks up to Week 48
Population: PK Population. Data for this endpoint was not collected as this study was terminated early during Part 1 as the risk benefit in relapsed/refractory AML did not favor continuation of the study.
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

38. Secondary Outcome: Part 2: Volume of Distribution of GSK2879552 for Part 2
Description: This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: as for outcome 37
Population: as for outcome 37
Groups:
- Part 2: Expansion Cohort: All Participants. Data for this endpoint was not collected as this study was terminated early during Part 1 as the risk benefit in relapsed/refractory AML did not favor continuation of the study.
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

39. Secondary Outcome: Number of Participants With Abnormal Covariates: Part 2
Description: This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: All Participants. Data for this endpoint was not collected as this study was terminated early during Part 1 as the risk benefit in relapsed/refractory AML did not favor continuation of the study.
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

40. Secondary Outcome: Duration of Response: Part 2
Description: This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 39
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

41. Secondary Outcome: Time to Time to Response: Part 2
Description: This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 39
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

42. Secondary Outcome: Progression-free Survival: Part 2
Description: This analysis was planned but not performed for Part 2 as the study was terminated early during Part 1.
Time Frame: Up to 14 months
Population: as for outcome 39
Arm/Group | Part 2: Expansion Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of the study up to 3 years
Description: All Treated Subjects Population was used to collect adverse events. AEs and SAEs were not collected in Part 2 of the study as no participants were enrolled due to early termination during Part 1.
Arm/Group | Part 1:GSK2879552 1mg QD | Part 1: GSK2879552 2mg QD | Part 1: GSK2879552 4mg QD | Part 1: GSK2879552 8mg QD | Part 1: GSK2879552 12mg QD | Part 1: GSK2879552 20mg QD | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day | Part 1: GSK2879552 20mg QD PK/PD Expansion | Part 2: Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 1/7 | 0/5 | 3/6 | 1/4 | 2/10 | 1/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 7/7 | 5/5 | 6/6 | 3/4 | 8/10 | 5/6 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 6/7 | 5/5 | 6/6 | 4/4 | 10/10 | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1:GSK2879552 1mg QD (N=1) | Part 1: GSK2879552 2mg QD (N=2) | Part 1: GSK2879552 4mg QD (N=7) | Part 1: GSK2879552 8mg QD (N=5) | Part 1: GSK2879552 12mg QD (N=6) | Part 1: GSK2879552 20mg QD (N=4) | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day (N=10) | Part 1: GSK2879552 20mg QD PK/PD Expansion (N=6) | Part 2: Expansion Cohort (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 2 (6) | 3 (5) | 3 (6) | 3 (3) | 1 (1) | 4 (4) | 3 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1:GSK2879552 1mg QD (N=1) | Part 1: GSK2879552 2mg QD (N=2) | Part 1: GSK2879552 4mg QD (N=7) | Part 1: GSK2879552 8mg QD (N=5) | Part 1: GSK2879552 12mg QD (N=6) | Part 1: GSK2879552 20mg QD (N=4) | Part 1: GSK2879552 2mg QD/ATRA 45mg/m^2/Day (N=10) | Part 1: GSK2879552 20mg QD PK/PD Expansion (N=6) | Part 2: Expansion Cohort (N=0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (6) | 3 (3) | 2 (4) | 1 (1) | 6 (6) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 4 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 4 (5) | 1 (4) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pseudohyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site vesicles (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arachnoid web (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 3 (4) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye haematoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT02177812/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT02177812/SAP_001.pdf